CLINICAL TRIAL: NCT02466126
Title: Effectiveness and Implementation of Brief Cognitive Behavioral Therapy in CBOCs
Acronym: MyBriefCBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 13-315
Record Dates: First submitted 2015-06-01; First posted 2015-06-09 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Depression
Keywords: Depression; brief Cognitive Behavioral Therapy (bCBT); Randomized Controlled Trial
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bCBT/Direct Referral (Experimental): A brief cognitive behavioral therapy intervention that offers 6 active- treatment sessions, each lasting 30 to 40 minutes, and telephone booster sessions to maintain changes.
  Interventions: Behavioral: bCBT
- Enhanced Usual Care (EUC) (No Intervention): Participants are provided with educational information on depression and will be encouraged to seek additional depression care options through their primary care providers.

INTERVENTIONS:
Behavioral: bCBT — The bCBT intervention uses 6 active-treatment sessions, each lasting 30 to 40 minutes, and telephone booster sessions to solidify changes. All participants receive an initial (core) session. In this session, participants work with their study clinician to set goals that are not restricted to "emotional health" (e.g., depression) but may also address "physical health" concerns (e.g., diet, exercise, managing a chronic condition). Following the core session, clinicians provide participants with a series of module choices, from which they select skills that match their most pressing needs. Each module focuses on a CBT technique (e.g., behavioral activation, changing thoughts), introduced and customized to the patient's immediate goals, regardless of the focus (physical or mental health).
  Arms: bCBT/Direct Referral

SUMMARY:
The purpose of this study is to determine the effectiveness of a brief cognitive behavioral therapy (bCBT) intervention for Veterans with depression delivered by mental health providers located at VA Community Based Outpatient Clinics (CBOC's) associated with the Houston and Oklahoma City VAMCs.

DETAILED DESCRIPTION:
Depression is a serious health condition that places tremendous burden on patients and healthcare systems and is especially prevalent in Veterans. In 2008, the VHA released the Uniform Mental Health Services Handbook (Handbook 1160.01) in an effort to expand services for Veterans with depression, including those in primary care and CBOC settings.

The VA remains a national leader in mental health services, but the provision of psychotherapy within VA is limited, especially for rural Veterans and those cared for in CBOCs. The VA has invested significant resources to improve access to high-quality mental health care, including a rapid expansion into CBOCs. Currently, there is a need to work with clinicians and stakeholders to address practice barriers related to mental health practices in CBOCs. A recent survey of 4,200 mental health providers in VA found that, although robust expansion and improved quality of mental health care services has occurred, access to proven effective psychotherapies in CBOCs remains a focused area for improvement. The study will examine whether existing VA CBOC mental health clinicians, with training and support, can effectively administer a structured brief cognitive behavioral therapy (bCBT) intervention for Veterans with clinically elevated symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

* must have clinically significant symptoms of depression;
* must be current recipients of services at CBOCs associated with the Houston and Oklahoma City VAMCs.

Exclusion Criteria:

* cognitive impairment;
* presence of bipolar, psychotic or substance-abuse disorders.
* Veterans currently receiving psychotherapy WILL be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Cully, PhD MEd, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (2):
- United States (2):
  - Oklahoma City VA Medical Center, Oklahoma City, OK, Oklahoma City, Oklahoma
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Johnson AL, Ecker AH, Fletcher TL, Hundt N, Kauth MR, Martin LA, Curran GM, Cully JA. Increasing the impact of randomized controlled trials: an example of a hybrid effectiveness-implementation design in psychotherapy research. Transl Behav Med. 2020 Aug 7;10(3):629-636. doi: 10.1093/tbm/iby116. PMID 30476315
- [Result] Brandt CP, Deavers F, Hundt NE, Fletcher TL, Cully JA. The Impact of Integrating Physical Health into a Brief CBT Approach for Medically Ill Veterans. J Clin Psychol Med Settings. 2020 Jun;27(2):285-294. doi: 10.1007/s10880-019-09634-2. PMID 31201653
- [Derived] Ecker AH, Shivaji S, Plasencia M, Kauth MR, Hundt NE, Fletcher TL, Sansgiry S, Cully JA. The role of symptom reduction in improving health-related quality of life through brief cognitive behavioral therapy. Psychother Res. 2025 Jul;35(6):972-980. doi: 10.1080/10503307.2024.2349992. Epub 2024 Jun 11. PMID 38861659
- [Derived] Rassu FS, Sansgiry S, Hundt NE, Kunik ME, Cully JA. Presence of PTSD is Associated with Clinical and Functional Impact in Veterans with Depression Treated in Community-Based Clinics. J Clin Psychol Med Settings. 2022 Mar;29(1):220-229. doi: 10.1007/s10880-021-09796-y. Epub 2021 Jun 22. PMID 34156589

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | bCBT/Direct Referral | Enhanced Usual Care (EUC)
Started | 109 | 80
Completed | 109 | 80
Not Completed | 0 | 0
Period: 4 Month Assessment
Arm/Group | bCBT/Direct Referral | Enhanced Usual Care (EUC)
Started | 109 | 80
Completed | 93 | 71
Not Completed | 16 | 9
Period: 8 Month Assessment
Arm/Group | bCBT/Direct Referral | Enhanced Usual Care (EUC)
Started | 93 | 71
Completed | 86 | 68
Not Completed | 7 | 3
Period: 12 Month Assessment
Arm/Group | bCBT/Direct Referral | Enhanced Usual Care (EUC)
Started | 86 | 68
Completed | 85 | 66
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | bCBT/Direct Referral | Enhanced Usual Care (EUC) | Total
Number analyzed (Participants) | 109 | 80 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (13.3) | 56.9 (13.8) | 58.3 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 102 | 69 | 171
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 68 | 55 | 123
  African American | 19 | 11 | 30
  American Indian/Alaskan Native | 6 | 1 | 7
  Asian/Vietnamese | 1 | 1 | 2
  Hispanic/Latino | 11 | 8 | 19
  Multiple Race | 4 | 3 | 7
  Unknown | 0 | 1 | 1
PHQ-9 [Count of Participants; unit: Participants] — The Patient Health Questionnaire (PHQ-9) is a measure used to access the level of depression a person is experiencing. Scores on the measure can range from 0 to 27. The higher the score the higher level of depression someone is experiencing. The measure was administered over the phone by an independent evaluator.
  Participants
    Moderate (10-14) | 37 | 32 | 69
    Moderate severe (15-19) | 47 | 28 | 75
    Severe (20-27) | 25 | 20 | 45
SF-12 [Mean (Standard Deviation); unit: units on a scale] — The SF-12V measures 8 concepts of health and can be summarized into summary component scores for physical (PCS) and mental (MCS) functioning. Scores can range from 0 - 100 and higher scores mean better functioning and quality of life. Population: The number of participants completing the assessment differs because some items were not completed by participants. If a participant didn't complete all of the items, then data was not used in the calculations.
  units on a scale
    SF - 12 PCS: number analyzed (Participants) | 106 | 77 | 183
    SF - 12 PCS | 33.12 (11.54) | 34.59 (13.12) | 33.74 (12.21)
    SF - 12 MCS: number analyzed (Participants) | 106 | 77 | 183
    SF - 12 MCS | 37.17 (9.79) | 34.43 (10.31) | 36.02 (10.07)
Beck Depression Inventory (BDI) [Mean (Standard Deviation); unit: units on a scale] — The measure will be used a s a second assessment to measure depression. Scores on the measure can range from 0 to 63. The higher the score the higher level of depression someone is experiencing. Population: The number of participants completing the assessment differs because some items were not completed by participants. If a participant didn't complete all of the items, then data was not used in the calculations.
  units on a scale
    number analyzed (Participants) | 99 | 68 | 167
    (all) | 25.65 (7.47) | 26.34 (8.33) | 25.93 (7.81)

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire (PHQ-9); Change in Depression Scores Taken at 4-, 8-, and 12-month Follow Ups as Compared to Baseline.
Description: The PHQ-9 is used to measure a person's level of depression. Scores on the measure can range from 0 to 27. The higher the score the higher level of depression someone is experiencing.
Time Frame: Baseline, 4-month (immediate post treatment), and 8- and 12-month follow up.
Population: The overall number of participants for each group was contacted to complete follow up assessments. Some participants declined to complete the assessment at each time point. Reasons for not completing assessments included: participants not interested in completing, unable to contact, and withdrew from the study. The population analyzed during the follow-up period represents the participants that agreed to complete the assessments for that time period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBT/Direct Referral | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 109 | 80
score on a scale
  Baseline | 16.40 (3.75) | 16.34 (4.24)
  4 Month: number analyzed (Participants) | 92 | 71
  4 Month | 11.74 (5.76) | 14.94 (5.51)
  8 Month: number analyzed (Participants) | 86 | 68
  8 Month | 12.79 (5.03) | 14.74 (5.67)
  12 Month: number analyzed (Participants) | 84 | 65
  12 Month | 12.99 (5.08) | 14.14 (5.40)

2. Secondary Outcome: Beck Depression Inventory (BDI) - Change is Being Assessed Using a 4 Timepoint Process
Description: The measure will be used a s a second assessment to measure depression. Scores on the measure can range from 0 to 63. The higher the score the higher level of depression someone is experiencing.
Time Frame: Baseline, 4-month (immediate post treatment), and 8- and 12-month follow up.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBT/Direct Referral | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 99 | 68
score on a scale
  Baseline | 25.65 (7.47) | 26.34 (8.33)
  4 Month: number analyzed (Participants) | 85 | 66
  4 Month | 18.98 (10.41) | 22.68 (10.07)
  8 Month: number analyzed (Participants) | 80 | 62
  8 Month | 20.23 (9.39) | 22.02 (10.89)
  12 Month: number analyzed (Participants) | 81 | 59
  12 Month | 20.72 (9.38) | 22.86 (10.99)

3. Secondary Outcome: Health Survey for Veterans (SF-12) - Change is Being Assessed Using a 4 Timepoint Process
Description: SF-12 will be used to measure a participant's functional status. The SF-12V measures 8 concepts of health and can be summarized into summary component scores for physical (PCS) and mental (MCS) functioning. Scores can range from 0 - 100 and higher scores mean better functioning and quality of life.
Time Frame: Baseline, 4-month (immediate post treatment), and 8- and 12-month follow up.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bCBT/Direct Referral | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 106 | 77
score on a scale
  Baseline: Physical Health | 33.12 (11.54) | 34.59 (13.12)
  Baseline: Mental Health | 37.17 (9.79) | 34.43 (10.31)
  4 Month: Physical Health: number analyzed (Participants) | 91 | 71
  4 Month: Physical Health | 31.46 (10.05) | 32.83 (12.21)
  4 Month: Mental Health: number analyzed (Participants) | 91 | 71
  4 Month: Mental Health | 41.84 (12.58) | 36.82 (10.03)
  8 Month: Physical Health: number analyzed (Participants) | 86 | 63
  8 Month: Physical Health | 29.72 (10.25) | 31.66 (12.05)
  8 Month: Mental Health: number analyzed (Participants) | 86 | 63
  8 Month: Mental Health | 39.76 (11.38) | 35.44 (11.37)
  12 Month: Physical Health: number analyzed (Participants) | 81 | 61
  12 Month: Physical Health | 30.98 (10.91) | 31.01 (11.87)
  12 Month: Mental Health: number analyzed (Participants) | 81 | 61
  12 Month: Mental Health | 38.41 (10.89) | 36.13 (11.27)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for a 12 month period.
Arm/Group | bCBT/Direct Referral | Enhanced Usual Care (EUC)
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/80
Other Adverse Events (participants affected / at risk) | 0/109 | 0/80

LIMITATIONS AND CAVEATS:
Study recruitment was hampered by a natural event, Hurricane Harvey. The event significantly slowed recruitment as part of the impact of the storm which hit the Houston area in August of 2017. The overall recruitment number was decreased to offset the better than expected retention of Veterans in the study. Re-calculated power analyses indicated that with our improved retention rates the study would require 189 Veteran participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT02466126/Prot_SAP_001.pdf